CLINICAL TRIAL: NCT00027521
Title: Phase I Study: Electroporation Therapy With Bleomycin For The Treatment Of Pancreatic Cancer
Brief Title: Electroporation Therapy With Bleomycin in Treating Patients With Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Program terminated
Sponsor: Ichor Medical Systems Incorporated (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069037; ICHOR-MCC-12305; MCC-12305; MCC-IRB-5948; NCI-V01-1672
Record Dates: First submitted 2001-12-07; First posted 2003-11-21 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bleomycin; Electroporation Therapies

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: electroporation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Electroporation therapy may enhance the ability of chemotherapy drugs to enter tumor cells. Combining chemotherapy with electroporation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of electroporation therapy and bleomycin in treating patients who have locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and surgical feasibility of electroporation therapy with bleomycin in patients with locally advanced pancreatic cancer. II. Determine the overall and progression-free survival of patients treated with this regimen.

OUTLINE: Patients receive bleomycin intratumorally during laparotomy. Approximately 15 minutes after the intratumoral injection, patients receive bleomycin IV over 10 minutes. Approximately 5 minutes after the IV injection, patients undergo electroporation therapy comprising electrical pulses directly to the pancreas and surrounding tissues. Patients are followed weekly for 4-6 weeks and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of adenocarcinoma of the pancreas Unresectable disease by exploratory laparotomy Involvement of the superior mesenteric artery or occlusion of the superior mesenteric vein-portal vein confluence No extrapancreatic metastases by ultrasound, CT scan, or laparotomy Tumor must be accessible for direct injection of study drug and placement of electrode array

PATIENT CHARACTERISTICS: Age: Any age Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: AST and ALT no greater than 3 times upper limit of normal No impaired hepatic function Renal: Creatinine no greater than 1.5 mg/dL No impaired renal function Cardiovascular: No impaired cardiac function Pulmonary: No compromised pulmonary function No pulmonary condition that would potentially require the use of high FIO2 levels Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study No prior reaction to bleomycin No fever, infection, or other medical condition that would preclude study Not at high risk for complications associated with abdominal surgery

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior lifetime cumulative dose of bleomycin greater than 400 U Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-12

CONTACTS AND LOCATIONS:
Overall Officials: Richard C. Karl, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute